CLINICAL TRIAL: NCT01952405
Title: Efficacy of Dialectical Behavior Therapy in Patients With Borderline Personality Disorder: a Controlled Trial in Taiwan
Brief Title: Efficacy of Dialectical Behavior Therapy in Patients With Borderline Personality Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Shen-Ing,Liu, Senior Visiting Staff, Mackay Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSC102-2314-B-195-002-My3
Record Dates: First submitted 2013-09-06; First posted 2013-09-30 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialectical behavior therapy (Experimental): Dialectical behavior therapy (DBT), developed by Marsha Linehan, has gained widespread popularity as a treatment for BPD, and its efficacy has been demonstrated in several trials.
  Interventions: Behavioral: Dialectical behavior therapy (DBT)
- alternative psychotherapy (Placebo Comparator): The therapists of the alternative psychotherapy in the comparison group are asked to provide the type and dose of therapy that they believed is most suited to the patient, with a minimum of 1 scheduled individual session per week. Ancillary treatment could be prescribed as needed. Case management strategies are also available in the comparison group (alternative psychotherapy group). No restrictions are placed on ancillary pharmacotherapy in either condition.
  Interventions: Behavioral: Dialectical behavior therapy (DBT)

INTERVENTIONS:
Behavioral: Dialectical behavior therapy (DBT) — Dialectical behavior therapy (DBT), developed by Marsha Linehan, has gained widespread popularity as a treatment for BPD, and its efficacy has been demonstrated in several trials.

SUMMARY:
The purpose of this study is to test the hypothesis:

Primary hypothesis: Participants in the dialectical behavior therapy group have greater reductions in the frequency and severity of suicidal and non-suicidal self-injurious behaviors compared to participants in the alternative treatment group.

Secondary Hypotheses: Participants in dialectical behavior therapy group have improved treatment outcomes compared to participants in alternative treatment, including mental health service utilization, symptoms of borderline personality and depression symptoms, suicidal thought and hopelessness, disability, and quality of life.

DETAILED DESCRIPTION:
This study will be a 3-year randomized control trial. Patients will be referred from any mental health services in Taipei area who meet Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision criteria for Borderline Personality Disorder. Inclusion criteria include subjects who fulfill the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision criteria for Borderline Personality Disorder, 18-60 years of age, sign the informed consent, have had at least two episodes of suicidal or non-suicidal self-injurious episodes in the past 5 years, and at least one of which is in the 3 months preceding enrollment. The exclusion criteria include psychotic disorder, bipolar I disorder, severe physical illness, and mental retardation. Outcome measures will be obtained at pre-treatment, 4-month, 8-month and post-treatment (12-month) during 1-year protocol. Using semi-structured interview and a battery of self-report forms, a range of symptoms and behaviors associated with Borderline Personality Disorder will be assessed including suicidal thought, suicide attempt, depression, hopelessness, quality of life, disability, service utilization, and function. Measures are selected based on previous outcome studies of dialectical behavior therapy. Outcome variables will be evaluated by blinded assessors.

ELIGIBILITY:
Inclusion Criteria:

* meeting DSM-IV criteria for borderline personality disorder
* 18-60 years of age
* have had at least two episodes of suicidal or non-suicidal self-injurious episodes in the past 5 years,
* at least one episode of suicidal is in the 3 months preceding enrollment
* agreement to participate in evaluation of the program.

Exclusion Criteria:

* bipolar I disorder, delirium, dementia, mental retardation, or a diagnosis of substance dependence in the preceding 30 days
* living outside of Taipei area
* having any serious medical condition likely to require hospitalization within the next year (e.g. cancer)
* and having plans to leave the Taipei area in the next 1 year

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05-18 (Actual); Primary Completion 2017-02-24 (Actual); Study Completion 2017-02-24 (Actual)

PRIMARY OUTCOMES:
Suicide Attempt Self-Injury Interview (SASII) | 4 months, 8 months and 12 months
  change from baseline in Suicide Attempt Self-Injury Interview at 4 months, 8 months and 12 months

SECONDARY OUTCOMES:
Borderline Personality Disorder Subscale | 4 months, 8 months and 12 months
  Borderline Personality Disorder Subscale (Chinese version) of the Structured Clinical Interview for DSM-IV axis II Personality Disorders ((SCID-II)
Borderline Symptom Checklist (BSL-23) | 4 months, 8 months and 12 months
The Patient Health Questionnaire (PHQ-9) | 4 months, 8 months and 12 months
Symptom Checklist-90-Revised (SCL-90-R) | 4 months , 8 months and 12 months
Beck Scale for Suicide Ideation (BSSI) | 4 months , 8months and 12 months
Beck Hopelessness Scale (BHS) | 4 months, 8 months and 12months
Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form (Q-LES-Q SF) | 4 months, 8 months and 12 months
Clinical Global Impressions-Severity (CGI-S) and Improvement (CGI-I) | 4 months, 8 months and 12 months
Brief Disability Questionnaire (BDQ) | 4 months, 8 months and 12 months
Treatment History Interview (THI) | 4 months, 8 months and 12 months

OTHER OUTCOMES:
The SCAN (Schedules for Clinical Assessment in Neuropsychiatry) | baseline assessment(0 month) and post-treatment (12-month)

CONTACTS AND LOCATIONS:
Overall Officials: Chie Pein Chen, PHD, Study Director — Department of Medical Research, Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: Click here for more information about this study — http://grbsearch.stpi.narl.org.tw/GRB/quickSearch.jsp